CLINICAL TRIAL: NCT03760939
Title: Clinical and Economical Evaluation of Colorectal Surgery in Ambulatory Care
Acronym: Colon-Ambu
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inclusion difficulties
Sponsor: IHU Strasbourg (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 18-001
Record Dates: First submitted 2018-11-29; First posted 2018-12-03 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Colorectal Surgery
Keywords: Colorectal surgery; Ambulatory care; Medical and economic evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ambulatory care (Experimental): Colorectal surgery in ambulatory care
  Interventions: Other: Clinical and economical evaluation
- Standard hospitalization (Other): Colorectal surgery with standard hospitalization for retrospective patients who benefit from the ERAS program, selected by statistical matching.
  Interventions: Other: Clinical and economical evaluation

INTERVENTIONS:
Other: Clinical and economical evaluation — Evaluation of the clinical and the economical impact of a colorectal surgery

SUMMARY:
Enhanced recovery after surgery (ERAS) significantly decreases mortality, morbidity and hospital length of stay without increasing the rate of re-hospitalization. It reduces psychologic stress caused by surgery and decreases postoperative complications about 50 %, especially in colorectal surgery. ERAS is now the object of several Good Practices Recommendations and is about to become the reference strategy.

The development of ambulatory surgery is a French national concern. Its interest has been demonstrated in many surgical fields. It requires a reflection centered on the patient and a health care pathway organization involving all health care actors.

While hospitalization is still the standard practice for colonic surgery, the objective of this study is to evaluate the medical and economic impact of an ambulatory care for colorectal surgery.

Ambulatory care will be compared to standard hospitalization of patients who benefit from the ERAS program.

DETAILED DESCRIPTION:
Enhanced recovery after surgery (ERAS) significantly decreases mortality, morbidity and hospital length of stay without increasing the rate of re-hospitalization. It reduces psychologic stress caused by surgery and decreases postoperative complications about 50 %, especially in colorectal surgery. ERAS is now the object of several Good Practices Recommendations and is about to become the reference strategy.

The development of ambulatory surgery is a French national concern. Its interest has been demonstrated in many surgical fields. It requires a reflection centered on the patient and a health care pathway organization involving all health care actors. Multiple interests have been shown:

* Equivalent mortality and/or morbidity compared with standard hospitalizations
* Medical and psychological benefits
* Individualized and less invasive health care pathways, in favor of patient's autonomy
* Multidisciplinary approach and innovative care
* Heath care costs management (decrease of hospital length of stay, optimization of operating rooms).

Ambulatory colectomies feasibility is recognized since 2013-2014 in France (Dr. Gignoux, MD in Lyon and Dr. Chasserant, MD in Le Havre). These ambulatory procedures are implemented in few expert centers with significant experience (more than 100 patients in Le Havre and more than 85 patients in Lyon) but several human and organizational limitations slow this innovative care.

The risk of complications does not seem to be increased on condition of anticipate and provide a postoperative follow-up at home.

While hospitalization is still the standard practice for colonic surgery, the objective of this study is to evaluate the medical and economic impact of an ambulatory care for colorectal surgery.

Ambulatory care will be compared to standard hospitalization of patients who benefit from the ERAS program.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 18 years old
* Patient able to understand the objectives and risks related to the trial
* Patient able to give written informed consent
* Patient able to understand and accept the health care program
* Isolated colonic lesion located on the colon or the upper rectum
* Any neoplastic or non-neoplastic colonic pathology
* Colonic surgery except resection without continuity interruption (e.g. low cecum resection, partial colectomy, suture for polyp)
* Moderate and/or controlled comorbidities
* No history of multiple laparotomies
* No psychosocial distress
* No living alone patient
* Patient registered with the French social security

Exclusion Criteria:

* Patient in exclusion period of another clinical study
* Emergency surgical procedure
* Type 1 diabetes
* Presence of an uncontrolled preoperative anemia
* Effective anticoagulation treatment, impossible to suspend
* Kidney failure (treated by dialysis)
* Hepatic cirrhosis
* Patient refusal
* Patient in custody
* Patient under guardianship
* Pregnancy
* Breastfeeding
* Poor general condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Mean cost evaluation | 1 month
  Mean cost evaluation, for the hospital, of the ambulatory care compared with standard hospitalization for patients who benefit from the ERAS program.

SECONDARY OUTCOMES:
Quality of life evaluation: EQ-5D (EuroQoL-5 Dimensions) scale | 7 and 30 days
  The EQ-5D Quality of Life scale consists of :
  (i) a descriptive system, consists in 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, extreme problems.
  (ii) a visual analog scale, records the respondent's self-rated health on a vertical, visual analogue scale where the endpoints are labelled 'Best imaginable health state" and "Worst imaginable health state".
Mean hospital length of stay | 2 years and 3 months
  Mean hospital length of stay for the "standard hospitalization" group
Ambulatory colectomies rate | 2 years and 3 months
  Rate of ambulatory colectomies compared to the total number of colectomies performed
Ambulatory care failure rate | 2 years and 3 months
  Rate of patients scheduled for ambulatory care and non-discharged the evening of surgery
Duty desk call | 2 years and 3 months
  Number of patients who called the duty desk (or for whom the duty desk has been called)
Mean time period required for a postoperative complication care | 2 years and 3 months
  Mean time period required for a postoperative complication care
Hospital re-admissions rate | 30 days
  Rate of hospital re-admissions related to postoperative complications
Rate of complications (Morbidity) | 30 days
  Rate of complications related or not to surgery
Rate of death (Mortality) | 30 days
  Number of patients who died within the individual participation period
Complications rate | 30 days
  Clinical and economic evaluation of postoperative complications rates difference between "ambulatory care" group and "standard hospitalization" group
Complications severity classification | 30 days
  Clinical and economic evaluation of complications severity assessed by the Clavien-Dindo classification
Evaluation of complication severity according to Clavien classification | 2 years and 3 months
  Severity of the complications will be evaluated according to the Clavien classification from Grade I "Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions" to Grade V "Death of a patient"
Mean additional hospital length of stay | 2 years and 3 months
  Clinical and economic evaluation of hospital length of stay related to complications difference between "ambulatory care" group and "standard hospitalization" group (additional hospitalizations, extension of hospitalization or new hospitalization).
Costs related to postoperative complications | 2 years and 3 months
  Costs related to postoperative complications difference between "ambulatory care" group and "standard hospitalization" group
Costs related to the management of postoperative complications | 2 years and 3 months
  Overall costs are evaluated by individual costs of:
  * unscheduled consultations,
  * surgical treatment,
  * medicated treatment
  * hospitalisation's duration

CONTACTS AND LOCATIONS:
Overall Officials: Didier Mutter, MD, PhD, Principal Investigator — Service Chirurgie Digestive et Endocrinienne, Nouvel Hôpital Civil de Strasbourg
Locations (1):
- Service de Chirurgie Digestive et Endocrinienne - Nouvel Hôpital Civil, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gignoux B, Pasquer A, Vulliez A, Lanz T. Outpatient colectomy within an enhanced recovery program. J Visc Surg. 2015 Feb;152(1):11-5. doi: 10.1016/j.jviscsurg.2014.12.004. Epub 2015 Feb 7. PMID 25661787
- [Background] Chasserant P, Gosgnach M. Improvement of peri-operative patient management to enable outpatient colectomy. J Visc Surg. 2016 Nov;153(5):333-337. doi: 10.1016/j.jviscsurg.2016.07.006. Epub 2016 Sep 23. PMID 27671006
- [Background] Slim K; Groupe GRACE (Groupe francophone de rehabilitation amelioree apres chirurgie); Amalberti R. Ambulatory colectomy: no innovation without evaluation. J Visc Surg. 2015 Feb;152(1):1-3. doi: 10.1016/j.jviscsurg.2015.01.001. Epub 2015 Jan 31. No abstract available. PMID 25650365
- [Background] Wind J, Polle SW, Fung Kon Jin PH, Dejong CH, von Meyenfeldt MF, Ubbink DT, Gouma DJ, Bemelman WA; Laparoscopy and/or Fast Track Multimodal Management Versus Standard Care (LAFA) Study Group; Enhanced Recovery after Surgery (ERAS) Group. Systematic review of enhanced recovery programmes in colonic surgery. Br J Surg. 2006 Jul;93(7):800-9. doi: 10.1002/bjs.5384. PMID 16775831
- [Background] Walter CJ, Collin J, Dumville JC, Drew PJ, Monson JR. Enhanced recovery in colorectal resections: a systematic review and meta-analysis. Colorectal Dis. 2009 May;11(4):344-53. doi: 10.1111/j.1463-1318.2009.01789.x. Epub 2009 Feb 4. PMID 19207699
- [Background] Gouvas N, Tan E, Windsor A, Xynos E, Tekkis PP. Fast-track vs standard care in colorectal surgery: a meta-analysis update. Int J Colorectal Dis. 2009 Oct;24(10):1119-31. doi: 10.1007/s00384-009-0703-5. Epub 2009 May 5. PMID 19415308
- [Background] Varadhan KK, Neal KR, Dejong CH, Fearon KC, Ljungqvist O, Lobo DN. The enhanced recovery after surgery (ERAS) pathway for patients undergoing major elective open colorectal surgery: a meta-analysis of randomized controlled trials. Clin Nutr. 2010 Aug;29(4):434-40. doi: 10.1016/j.clnu.2010.01.004. Epub 2010 Jan 29. PMID 20116145
- [Background] Adamina M, Kehlet H, Tomlinson GA, Senagore AJ, Delaney CP. Enhanced recovery pathways optimize health outcomes and resource utilization: a meta-analysis of randomized controlled trials in colorectal surgery. Surgery. 2011 Jun;149(6):830-40. doi: 10.1016/j.surg.2010.11.003. Epub 2011 Jan 14. PMID 21236454
- [Background] Spanjersberg WR, Reurings J, Keus F, van Laarhoven CJ. Fast track surgery versus conventional recovery strategies for colorectal surgery. Cochrane Database Syst Rev. 2011 Feb 16;(2):CD007635. doi: 10.1002/14651858.CD007635.pub2. PMID 21328298
- [Background] Slim K, Delaunay L, Joris J, Leonard D, Raspado O, Chambrier C, Ostermann S; Le Groupe francophone de rehabilitation amelioree apres chirurgie (GRACE). How to implement an enhanced recovery program? Proposals from the Francophone Group for enhanced recovery after surgery (GRACE). J Visc Surg. 2016 Dec;153(6S):S45-S49. doi: 10.1016/j.jviscsurg.2016.05.008. Epub 2016 Jun 14. No abstract available. PMID 27316295
- [Background] Gustafsson UO, Oppelstrup H, Thorell A, Nygren J, Ljungqvist O. Adherence to the ERAS protocol is Associated with 5-Year Survival After Colorectal Cancer Surgery: A Retrospective Cohort Study. World J Surg. 2016 Jul;40(7):1741-7. doi: 10.1007/s00268-016-3460-y. PMID 26913728
- [Background] Lawrence JK, Keller DS, Samia H, Ermlich B, Brady KM, Nobel T, Stein SL, Delaney CP. Discharge within 24 to 72 hours of colorectal surgery is associated with low readmission rates when using Enhanced Recovery Pathways. J Am Coll Surg. 2013 Mar;216(3):390-4. doi: 10.1016/j.jamcollsurg.2012.12.014. Epub 2013 Jan 23. PMID 23352608
- [Background] Bardram L, Funch-Jensen P, Jensen P, Crawford ME, Kehlet H. Recovery after laparoscopic colonic surgery with epidural analgesia, and early oral nutrition and mobilisation. Lancet. 1995 Mar 25;345(8952):763-4. doi: 10.1016/s0140-6736(95)90643-6. PMID 7891489
- [Background] Levy BF, Scott MJ, Fawcett WJ, Rockall TA. 23-hour-stay laparoscopic colectomy. Dis Colon Rectum. 2009 Jul;52(7):1239-43. doi: 10.1007/DCR.0b013e3181a0b32d. PMID 19571699
- [Background] Gash KJ, Goede AC, Chambers W, Greenslade GL, Dixon AR. Laparoendoscopic single-site surgery is feasible in complex colorectal resections and could enable day case colectomy. Surg Endosc. 2011 Mar;25(3):835-40. doi: 10.1007/s00464-010-1275-8. Epub 2010 Aug 24. PMID 20734083
- [Background] Rogers JP, Dobradin A, Kar PM, Alam SE. Overnight hospital stay after colon surgery for adenocarcinoma. JSLS. 2012 Apr-Jun;16(2):333-6. doi: 10.4293/108680812x13427982376789. PMID 23477191
- [Background] Dobradin A, Ganji M, Alam SE, Kar PM. Laparoscopic colon resections with discharge less than 24 hours. JSLS. 2013 Apr-Jun;17(2):198-203. doi: 10.4293/108680813X13654754535791. PMID 23925012
- [Background] Martin-Ferrero MA, Faour-Martin O, Simon-Perez C, Perez-Herrero M, de Pedro-Moro JA. Ambulatory surgery in orthopedics: experience of over 10,000 patients. J Orthop Sci. 2014 Mar;19(2):332-338. doi: 10.1007/s00776-013-0501-3. Epub 2014 Jan 7. PMID 24395115
- [Background] Verrier JF, Paget C, Perlier F, Demesmay F. How to introduce a program of Enhanced Recovery after Surgery? The experience of the CAPIO group. J Visc Surg. 2016 Dec;153(6S):S33-S39. doi: 10.1016/j.jviscsurg.2016.10.001. Epub 2016 Nov 16. PMID 27863944
- [Background] Daams F, Wu Z, Lahaye MJ, Jeekel J, Lange JF. Prediction and diagnosis of colorectal anastomotic leakage: A systematic review of literature. World J Gastrointest Surg. 2014 Feb 27;6(2):14-26. doi: 10.4240/wjgs.v6.i2.14. PMID 24600507
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542